CLINICAL TRIAL: NCT00902707
Title: An Open-Label, 2-way Crossover Placebo-Controlled , Radio-Labeled Tracer Study Evaluating the Effect of MUCINEX® 1200 mg on Mucociliary and Cough Clearance From The Human Lung In Healthy, Non-Smoking Adults
Brief Title: Evaluating the Effect of Mucinex® 1200 mg on Mucociliary and Cough Clearance From the Human Lung
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Reckitt Benckiser Inc. (Industry)
Responsible Party: Principal Investigator, William Bennett, PhD, Professor of Medicine, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-MUC-01
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-05

CONDITIONS: Mucociliary Clearance
Keywords: healthy nonsmokers
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mucinex 1200mg (Experimental): Pill
  Interventions: Drug: Mucinex 1200mg
- Placebo (Placebo Comparator): Pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mucinex 1200mg — Compared to Placebo
  Arms: Mucinex 1200mg
Drug: Placebo — Compare to active Mucinex
  Arms: Placebo

SUMMARY:
The purpose of this research study is to test the ability of Mucinex, an oral, over-the-counter, FDA approved expectorant) to stimulate the clearance of inhaled particles from the subject's lungs (called "mucociliary clearance"). The study will also monitor the metabolism of the drug by the subject's body.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non smoker
* BMI 19-29
* Normal lung function

Exclusion Criteria:

* Pregnant
* Smokers
* Any illness

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Difference between drug and placebo in the percentage of particles cleared from the lung. | Measurements at 60, 90 and 180 min
Difference between drug and placebo as an estimate of small airway clearance. | Measurements at 60, 90 and 180 min
Difference between drug and placebo between study days. | Measurements at 60, 90 and 180 min

SECONDARY OUTCOMES:
Blood will be drawn to determination of guaifenesin in the serum. | at baseline and every 30 min x8

CONTACTS AND LOCATIONS:
Overall Officials: William Bennett, PhD, Principal Investigator — University of North Carolina
Locations (1):
- UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States